CLINICAL TRIAL: NCT05515289
Title: Study of SHR6390 in Renal Insufficiency and Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SHR6390-I-114
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — dalpiciclib

STUDY DESIGN:
Intervention Model Description: The study is a single-center, open, single-dose, self-controlled clinical trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group: mild renal insufficiency (Experimental)
  Interventions: Drug: SHR6390
- Treatment group: moderate renal insufficiency (Experimental)
  Interventions: Drug: SHR6390
- Treatment group: healthy subjects (Experimental)
  Interventions: Drug: SHR6390

INTERVENTIONS:
Drug: SHR6390 — SHR6390 tablet single dose, and subjects will take the SHR6390 on Day 1.
  Other Names: dalpiciclib

SUMMARY:
The study is a single-center, open, single-dose, self-controlled clinical trial. It is planned to enroll 24-30 subjects.

Subjects will take the SHR6390 on Day1.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with renal insufficiency

1. Sign an informed consent form before the test, and fully understand the content, process and possible adverse reactions of the test;
2. Age 18 to 70 years old, gender is not limited;
3. Body mass index (BMI) in the range of 19 kg/m2 to 28 kg/m2 (including both ends);
4. Renal function index (expressed in GFR, by the MDRD formula (refer to Appendix I) meets the following criteria: Subjects with mild renal insufficiency (stage CKD2): 60-89 mL/min (both ends included)；Subjects with moderate renal insufficiency (stage CKD3): 30-59 mL/min (both ends included)；
5. The renal function state is stable, and the GFR results of the two tests before administration (the interval between the two tests should be at least 3 days) should be within the same CKD segmentation period;
6. Fertile female subjects must undergo a pregnancy test before administration and the result is negative; must be non-lactating; Female subjects with fertility who used medically approved, highly effective contraception for 7 months from the signing of informed consent to the last dose; Male subjects whose partners are fertile women, who use medically approved, highly effective contraception for 4 months after the last dose; There are no sperm donations, egg donations and fertility plans.

Healthy subjects

1. Sign an informed consent form before the test, and fully understand the content, process and possible adverse reactions of the test;
2. Age 18 to 70 years old, gender is not limited;
3. Body mass index (BMI) in the range of 19 kg/m2 to 28 kg/m2 (including both ends);
4. Renal function index (expressed in GFR, calculated as above) ≥ 90 mL/min and < 130 mL/min;
5. Comprehensive vital signs examination, physical examination, routine laboratory examination (blood routine, blood biochemistry, urine routine, coagulation function, etc.), 12-lead ELECTROCardiogram, X-chest x-ray or chest CT, abdominal ultrasound and other examinations have been judged by the researchers to be normal or abnormal and have no clinical significance;
6. The principle of gender ratio matching in the health group: try to match the sex ratio of men and women in the renal insufficiency group; The age matching principle is: ± 10 years old; The fasting weight matching principle is: ± 10 kg;
7. Fertile female subjects must undergo a pregnancy test before administration and the result is negative; must be non-lactating; Female subjects with fertility who used medically approved, highly effective contraception for 7 months from the signing of informed consent to the last dose; Male subjects whose partners are fertile women, who use medically approved, highly effective contraception for 4 months after the last dose; There are no sperm donations, egg donations and fertility plans. (Refer to Appendix II).

Exclusion Criteria:

- Subjects with renal insufficiency

1. Have had a kidney transplant;
2. Renal dialysis is required during the study;
3. Urinary incontinence or anuresis;
4. People who are allergic to research drugs or excipients;
5. Clinically significant heart disease within 12 months prior to the start of treatment, including but not limited to: congestive heart failure, symptomatic coronary artery disease, arrhythmia, myocardial infarction, QTcF≥470 ms (female) or 450 ms (male), etc.;
6. Coagulation dysfunction (INR>1.5) or prothrombin time (PT) >ULN + 4 seconds or APTT >1.5 ×ULN), or clinically significant bleeding symptoms or clear bleeding tendencies within 3 months before screening, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, etc., or receiving thrombolytic anticoagulation;
7. Laboratory tests such as blood routine and blood biochemistry show that the functional level of the organ meets the following abnormalities (no blood transfusion or hematopoietic growth factor therapy is received within 2 weeks before the blood routine screening):

   * Neutrophil absolute values < 1.5×109/L；
   * Absolute lymphocyte value < 0.8×109/L ;
   * Platelet count <150×109/L；
   * Total bilirubin > 1.5 × ULN;
   * ALT and AST>2×ULN;
8. Patients with hypertension who cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥90 mmHg);
9. Liver diseases that affect metabolism or digestive tract diseases that affect absorption;
10. Those who donated 400 mL of blood ≥ in the 3 months before screening, or 200 mL ≥ 1 month before screening, or who received blood transfusions;
11. Screening of those who have used any clinical trial drugs in the previous 3 months;
12. Drugs that induce CYP3A, CYP2C8, CYP2C9 enzymes were used 28 days before taking the study drug, and drugs with inhibitory effects on CYP3A, CYP2C8, CYP2C9 enzymes were used 14 days before taking the study drug, or needed to be used during the trial, any drug that affects the metabolic enzymes CYP3A, CYP2C8, CYP2C9; or use any Chinese medicine or proprietary Chinese medicine 7 days before taking the research drug;
13. Alcoholics (drink 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine; 5 cigarettes smoked per day≥), or those who could not smoke and abstain from alcohol during the trial period, or those who screened positive for alcohol;
14. Those who have a positive urine drug abuse screening, or those who have a history of drug abuse in the past five years or who have used drugs in the 3 months before the test;
15. Active HBV infection (gene copy number test for HBsAg positive), or positive for HCV and syphilis antibodies;
16. Have a history of immunodeficiency (including HIV test-positive, other acquired, congenital immunodeficiency diseases) or organ transplantation;
17. 48 hours before taking the study drug until the end of the study, subjects refused to stop any beverage containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or grapefruit (grapefruit) or grapefruit and products containing grapefruit or grapefruit ingredients (grapefruit juice, grapefruit juice, etc.);
18. 48 hours before taking the drug until the end of the study, the subject exercised vigorously, or had other factors affecting the absorption, distribution, metabolism and excretion of the drug;
19. Those who were vaccinated live within 2 weeks prior to the first use of the study drug, or who planned to receive live vaccination within 7 days of the end of the study
20. Subjects who the investigator believes have other factors that are not suitable for participating in this test.

Healthy subjects

1. Have had a kidney transplant;
2. People who are allergic to research drugs or excipients;
3. Clinically significant heart disease within 12 months before the start of treatment, including but not limited to: congestive heart failure, symptomatic coronary artery disease, arrhythmia, myocardial infarction, QTcF≥470 ms (female) or 450 ms (male), etc.;
4. Coagulation dysfunction (INR>1.5) or prothrombin time (PT) >ULN +4 seconds or APTT >1.5 ×ULN), or clinically significant bleeding symptoms or clear bleeding tendencies such as gastrointestinal bleeding, hemorrhagic gastric ulcers, etc., within 3 months before screening, or receiving thrombolytic anticoagulation;
5. There is a clear medical history of primary diseases of important organs such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and skeletal musculoskeletal system, etc., and the researchers believe that they are not suitable for participating in this study;
6. Those who donated 400 mL of blood ≥ 3 months before screening, or 200 mL of blood donated in≥ 1 month before screening, or who received blood transfusions;
7. Screening of those who have used any clinical trial drugs in the previous 3 months;
8. Drugs that induce CYP3A, CYP2C8, CYP2C9 enzymes were used 28 days before taking the research drug, and drugs with inhibitory effect on CYP3A, CYP2C8, CYP2C9 enzymes were used 14 days before taking the research drug, or needed to be used during the trial, any drug that affects the metabolic enzymes CYP3A, CYP2C8, CYP2C9; or use any Chinese medicine or proprietary Chinese medicine 7 days before taking the research drug;
9. Alcoholics (drink 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine; 5 cigarettes smoked per day≥), or those who could not smoke and abstain from alcohol during the trial period, or those who screened positive for alcohol;
10. Urine drug abuse screening positive, or those who have a history of drug abuse in the past five years or have used drugs in the 3 months before the test;
11. Positive HBsAg, HCV or syphilis antibody test;
12. Have a history of immunodeficiency (including HIV test-positive, other acquired, congenital immunodeficiency diseases) or organ transplantation;
13. 48 hours before taking the study drug until the end of the study, the subject refused to stop any beverage containing methylxanthine, such as caffeine (coffee, tea, cola, chocolate, etc.) or alcoholic beverages or grapefruit (grapefruit) or grapefruit and products containing grapefruit or grapefruit ingredients (grapefruit juice, grapefruit juice, etc.);
14. 48 hours before taking the drug until the end of the study, the subject exercised vigorously, or had other factors affecting the absorption, distribution, metabolism and excretion of the drug;
15. Those who were vaccinated live within 2 weeks prior to the first use of the study drug, or who planned to be vaccinated within 7 days of the end of the study
16. Inability to receive a uniform diet and inability to tolerate indwelling needles for intravenous blood collection;
17. Subjects who the investigator believes have other factors that are not suitable for participating in this test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-08-28 (Estimated); Study Completion 2023-09-28 (Estimated)

PRIMARY OUTCOMES:
Dalpiciclib main pharmacokinetic parameters: Cmax | from Day 1 to Day 10
Dalpiciclib main pharmacokinetic parameters: AUC0-t | from Day 1 to Day 10
Dalpiciclib main pharmacokinetic parameters: AUC0-∞ | from Day 1 to Day 10

SECONDARY OUTCOMES:
Secondary pharmacokinetic parameters of Dalpiciclib: Tmax | from Day 1 to Day 10
Secondary pharmacokinetic parameters of Dalpiciclib: t1/2 | from Day 1 to Day 10
Secondary pharmacokinetic parameters of Dalpiciclib: CL/F | from Day 1 to Day 10
Secondary pharmacokinetic parameters of Dalpiciclib: Vz/F | from Day 1 to Day 10
Secondary pharmacokinetic parameters of Dalpiciclib: CLR | from Day 1 to Day 10
Secondary pharmacokinetic parameters of Dalpiciclib: Ae | from Day 1 to Day 10
Secondary pharmacokinetic parameters of Dalpiciclib: Ae% | from Day 1 to Day 10
Incidence and severity of good/serious adverse events (rated based on CTCAE v5.0) | from Day1 to Day19，an average of 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital Southesat University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided